CLINICAL TRIAL: NCT01766271
Title: GENErating Change, An Integrative Health Coaching and Genetic Risk Testing Pilot in Primary Care: A Multidisciplinary Approach to Personalized Medicine Targeting CHD Risk
Brief Title: GENErating Behavior Change, An Integrative Health Coaching and Genetic Risk Testing Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00029973
Record Dates: First submitted 2012-10-15; First posted 2013-01-11 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Heart Disease Risk
Keywords: Coronary heart disease; cardiovascular disease; risk
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Risk Assessment (SRA) Only (Experimental)
  Interventions: Other: Standard Risk Assessment
- SRA plus Health Coaching (Experimental)
  Interventions: Behavioral: Health Coaching; Other: Standard Risk Assessment
- SRA plus Genetic Testing (Experimental)
  Interventions: Genetic: 9p21; Other: Standard Risk Assessment
- SRA plus Health Coaching plus Genetic Testing (Experimental)
  Interventions: Behavioral: Health Coaching; Genetic: 9p21; Other: Standard Risk Assessment

INTERVENTIONS:
Behavioral: Health Coaching — biweekly health coaching for 5 months
  Arms: SRA plus Health Coaching; SRA plus Health Coaching plus Genetic Testing
Genetic: 9p21 — Genetic testing results of 9p21
  Arms: SRA plus Genetic Testing; SRA plus Health Coaching plus Genetic Testing
Other: Standard Risk Assessment — All 4 arms are assigned to receive standard assessment on coronary heart disease risk

SUMMARY:
The purpose of this 4 group (2x2) pilot randomized controlled trial is to test the feasibility and logistics of incorporating genetic risk information (9p21)into standard Coronary Heart Disease (CHD) risk counseling or health coaching intervention (or both) in primary care at 2 Duke Clinics.

ELIGIBILITY:
Inclusion Criteria:

* age 18+,
* presence of at least one of the following:

  * FPG > 100,
  * HbA1c > 5.7%,
  * diabetic,
  * LDL > 129,
  * triglycerides > 150,
  * total cholesterol > 200,
  * SBP > 130,
  * BMI > 25,
* able to speak and understand English,
* able and willing to give informed consent

Exclusion Criteria:

* diagnosed CHD (MI or documented coronary artery disease),
* inability to ambulate or participate in physical activity,
* serious chronic disease related complications,
* current participation in a risk communication study for chronic disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Diet | 6 months
  National Cancer Institute (NCI) Multifactor Screener
Physical Activity | 6 months
  Stanford Brief Activity Scale (SBAS)

SECONDARY OUTCOMES:
Fasting blood glucose | 6 months
Systolic blood pressure | 6 months
Body mass index | 6 months
Waist circumference | 6 months
Low Density Cholesterol (LDL) | 6 months
Triglyceride | 6 months
Total cholesterol | 6 months